CLINICAL TRIAL: NCT05106075
Title: Pilot Study to Validate ex Vivo Expression of Specific Biomarkers of Human Resolutive Macrophages
Acronym: RESOMACRO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2020/562
Record Dates: First submitted 2021-10-08; First posted 2021-11-03 (Actual); Last update posted 2021-11-03 (Actual); Status verified 2021-10

CONDITIONS: Inflammation
Keywords: macrophage; inflammation; inflammation resolution
MeSH Terms: conditions — Inflammation | interventions — Blood Specimen Collection

STUDY DESIGN:
Masking Description: patients are anonymized
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- biologic sample collection (Experimental): Blood samples or gingival exsudat collection
  Interventions: Procedure: blood sample or joint fluid or gingival exudate

INTERVENTIONS:
Procedure: blood sample or joint fluid or gingival exudate — blood sample collected by peripheral blood mobilization joint fluid collected by punction gingival exudate collected with paper strips

SUMMARY:
Human resolutive macrophages are essential immune cells in the resolution of inflammation. This particular type of macrophages remains poorly known and currently there are no biomarkers to identify them in vivo. Within UMR1098-RIGHT, specific biomarkers (secreted molecules and membrane receptors) of human resolutive macrophages (healthy volunteers) have been identified in vitro, but their existence in vivo remains an outstanding issue. An exploratory study (lack of data from the literature) will validate the ex vivo expression of these markers in samples of patients whose inflammation is not, or little, supported by the available therapies (NSAIDs, biotherapies, corticosteroids).

ELIGIBILITY:
Inclusion Criteria:

* Age Limits (18-80 years)
* Information and non-opposition for participating in the study
* Patients suffering from periodontitis grade III ou IV
* Patients suffering from microcristalline arthritis
* patient with health insurance

Exclusion Criteria:

* patient under corticotherapy
* pregnancy
* non-compliant patient
* patient with no health insurance
* patient in exclusion period from an other study
* legal incapacity

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-07-07 (Actual); Primary Completion 2024-01-07 (Estimated); Study Completion 2024-01-07 (Estimated)

PRIMARY OUTCOMES:
Quantification of cytokine concentrations in samples by ELISA | up to 2 months

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - CHRU Besançon, Besançon
  - Dentist'S Office, Montbéliard

IPD SHARING:
Plan to Share IPD: No